CLINICAL TRIAL: NCT04542408
Title: Hamburg Edoxaban for Anticoagulation in COVID-19 Study
Acronym: HERO-19
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Universitätsklinikum Hamburg-Eppendorf (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HERO-19
Record Dates: First submitted 2020-09-06; First posted 2020-09-09 (Actual); Last update posted 2023-05-23 (Actual); Status verified 2023-05

CONDITIONS: Covid19
Keywords: Coagulopathy
MeSH Terms: conditions — COVID-19; Hemostatic Disorders | interventions — Anticoagulants; edoxaban; Heparin, Low-Molecular-Weight

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intensive anticoagulation strategy (Experimental): In-hospital (ICU & normal ward): weight-adapted LMWH, high dose/ therapeutic dose (according to respective SmPC) After discharge and in ambulatory patients: Edoxaban according to SmPC
  Interventions: Drug: Anticoagulation Agents (Edoxaban and/or high dose LMWH)
- Moderate anticoagulation strategy (Other): In-hospital (ICU & normal ward): LMWH, prophylactic dose as part of SOC After discharge and in ambulatory patients: Administration of oral placebo according to the dosing rules for Edoxaban
  Interventions: Drug: Low dose Low molecular weight heparin or Placebo

INTERVENTIONS:
Drug: Anticoagulation Agents (Edoxaban and/or high dose LMWH) — In-hospital (ICU & normal ward): weight-adapted LMWH, high dose/ therapeutic dose (according to respective SmPC) After discharge and in ambulatory patients: Edoxaban according to SmPC until
  Arms: Intensive anticoagulation strategy
Drug: Low dose Low molecular weight heparin or Placebo — In-hospital (ICU & normal ward): LMWH, prophylactic dose as part of SOC After discharge and in ambulatory patients: Administration of oral pla-cebo according to the dosing rules for Edoxaban
  Arms: Moderate anticoagulation strategy

SUMMARY:
Hero-19 aims to evaluate if an intensive anticoagulation strategy using Edoxaban on top of standard of care (SOC) of COVID-19 therapy is superior to SOC (in-hospital moderate anticoagulation strategy = low-dose low-molecular weight heparin [LMWH], ambulatory no anticoagulation, i.e. placebo within this trial) in reduction of morbidity and mortality endpoints in patients with COVID-19.

DETAILED DESCRIPTION:
Coagulopathy in the context of COVID-19 is a major threat to affected patients due to deep vein thromboses and pulmonary embolisms. Actual data show an unexpectedly high incidence of partially fatal complications without any prior clinical evidence in some cases. Therefore, this prospective, randomized, assessor-blinded, multicenter, placebo-controlled, interventional trial will investigate whether therapeutic anticoagulation on top of SOC compared to prophylactic anticoagulation as part of SOC- can improve objective patient-relative endpoints, relevant for prognosis in patients with COVID-19. 172 eligible patients will be randomized 1:1 to experimental or control group. Patients enrolled to experimental group will receive therapeutic anticoagulation using LMWH body weight-adapted during course of hospital stay and oral anticoagulation using Edoxaban according to SmPC (60mg once a day) after being discharged from hospital / outpatient course. Patients enrolled to control group will receive prophylactic anticoagulation using LMWH as part of SOC whilst inpatient course, and placebo after discharge / outpatient course. Patients will be informed of their allocation to the placebo group, as it has been shown that the effect of placebo is still detectable.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of COVID-19 and hospitalization on ICU, or
* Diagnosis of COVID-19 and hospitalization on normal ward, or
* Diagnosis of COVID-19 (within 10 days) and troponin ≥ ULN and/or D-dimer ≥0.5 mg/L

Exclusion Criteria:

* Age below 18
* Life expectancy less than 3 months before COVID-19
* Resuscitation > 30 minutes
* Hypersensitivity to the active substance, to Edoxaban or any of its excipients
* Significantly increased bleeding risk
* Other indication for anticoagulation beyond COVID-19
* GFR < 15 ml/min
* Planned transfer of the patient to another clinic within the next 42 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2020-11-12 (Actual); Primary Completion 2022-09-06 (Actual); Study Completion 2023-01-15 (Actual)

PRIMARY OUTCOMES:
Combined endpoint: all-cause mortality and/ or venous thromboem-bolism and/ or arterial thromboembolism | 42 days
  All-cause mortality and/ or venous thromboem-bolism and/ or arterial thromboembolism during follow-up (42 days). Thromboembolisms will be detected by duplex ultrasonography of arms and legs.

SECONDARY OUTCOMES:
All-cause mortality | 42 days
  All-cause mortality during follow-up (42 days)
Mortality related to venous thromboembolism | 42 days
  Mortality related to venous thromboembolism during follow-up (42 days)
Mortality related to arterial thromboembolism | 42 days
  Mortality related to arterial thromboembolism during follow-up (42 days)
Rate of venous and/ or arterial thromboembolism | 42 days
  Rate of venous and/ or arterial thromboembolism during follow-up (42 days) Thromboembolisms will be detected by duplex ultrasonography of arms and legs
Rate and length of mechanical ventilation | 42 days
  Rate and length of mechanical Ventilation during follow-up (42 days)
Length of initial stay at ICU after application of IMP | 42 days
  Length of initial stay at ICU after application of IMP during follow-up (42 days)
Rehospitalisation | 42 days
  Rehospitalisation during follow-up (42 days)
Rate and length of renal replacement therapy | 42 days
  Rate and length of renal replacement therapy during follow-up (42 days)
Cardiac arrest/ CPR | 42 days
  Cardiac arrest/ CPR during follow-up (42 days)

CONTACTS AND LOCATIONS:
Overall Officials: Stefan Kluge, MD, Principal Investigator — Universitätsklinikum Hamburg-Eppendorf
Locations (10):
- Germany (10):
  - UK Aachen, Aachen
  - Universitätsklinikum Augsburg, Augsburg
  - Universitätsklinikum Düsseldorf, Düsseldorf
  - Universitätsklinikum Freiburg, Freiburg im Breisgau
  - Asklepios Klinik Altona, Hamburg
  - Asklepios Klinik Barmbek, Hamburg
  - Asklepios Klinik St. Georg, Hamburg
  - Universitärsklinikum Hamburg-Eppendorf, Hamburg
  - Medizinische Hochschule Hannover, Hanover
  - TU München Klinikum rechts der Isar, München

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Santos BC, Flumignan RL, Civile VT, Atallah AN, Nakano LC. Prophylactic anticoagulants for non-hospitalised people with COVID-19. Cochrane Database Syst Rev. 2023 Aug 16;8(8):CD015102. doi: 10.1002/14651858.CD015102.pub2. PMID 37591523